CLINICAL TRIAL: NCT07368127
Title: A Single-Arm, Open-Label, Dose-Escalation/Cohort-Expansion Phase Ia/Ib Study to Evaluate Safety, Tolerability, PK/PD Profiles, and Preliminary Efficacy of TPD3310 Injection in Advanced Malignant Solid Tumor Patients
Brief Title: A Study of TPD3310 in Patients With Advanced Malignant Tumors
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: TAIBIDI PHARMACEUTICAL TECHNOLOGY(SHIJIAZHUANG) CO.,LTD. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TBD CA101
Record Dates: First submitted 2026-01-03; First posted 2026-01-26 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2025-12

CONDITIONS: Advanced Malignant Solid Tumors
Keywords: Neoplasms; Antineoplastic Agents
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TPD3310 monotherapy (Experimental): • Phase Ia: Single and Multiple Dose Escalation. • Phase Ib: Cohort Expansion.
  Interventions: Drug: TPD3310 injection

INTERVENTIONS:
Drug: TPD3310 injection — * Phase Ia: Single and Multiple Dose Escalation. (1) Dosage form: injection. (2) Dosage: 6 dose groups, 50 mg, 100 mg, 200 mg, 350 mg, 500 mg, 650 mg,.-Arms Assigned Interventions (3) Frequency: once weekly. (4) Duration: days 1-21; 28 days per cycle.
  * Phase Ib: Cohort Expansion. Dosage and dosing regimen: according to the recommended dosage and dosing cycle from the Phase Ia study.

SUMMARY:
This study is a multicenter, open phase I clinical study of dose escalation,cohort expansion study to evaluate the safety,tolerability,pharmacokinetics,pharmacodynamics, and preliminary efficacy of TPD3310 in patients withadvanced malignant solid tumors.

DETAILED DESCRIPTION:
TPD3310 is a selective c-MET degrader, and this is the first-in-human trial of TPD3310. This study adopts an open-label, non-randomized, single-arm, dose-escalation, and cohort expansion research design, and is divided into two parts, Phase Ia and Phase Ib.

Phase Ia is a single and multiple dose escalation trial with an open-label design, aiming to evaluate the safety, tolerability, PK, and PD characteristics of TPD3310 tablets, preliminarily assess the anti-tumor efficacy, and recommend the dose for Phase Ib study.

Phase Ib is a single-arm cohort expansion study conducted in participants with six solid tumors, based on the recommended dosage and dosing cycle from the Phase Ia study. The actual tumor types for the Phase Ib study will be adjusted according to the safety and efficacy data from the Phase Ia study.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily sign the informed consent form and follow protocol requirements.
2. Aged 18 to 75 (both inclusive), male or female, regardless of race.
3. Expected survival period ≥ 12 weeks.
4. ECOG PS score ≤1.
5. Phase Ia study:

   •Patients with pathologically or cytologically confirmed advanced malignant solid tumors (not limited to lung cancer, gastric cancer, liver cancer and cholangiocarcinoma, esophageal cancer, pancreatic cancer, and renal cancer) who have progressive disease despite standard treatment, are intolerant to standard treatment, or lack effective standard treatment; c-MET positive patients are preferred. At least one measurable lesion meeting RECIST v1.1 criteria;

   Phase Ib study:
   * Cohort A (histologically or cytologically confirmed lung cancer, failed or intolerant to standard treatment, EGFR wild-type, c-MET positive. Investigators may adjust enrollment criteria after communicating with the sponsor based on subjects' efficacy responses during the trial.), Cohort B (histologically or cytologically confirmed esophageal cancer, failed or intolerant to standard treatment, c-MET positive. Investigators may adjust enrollment criteria after communicating with the sponsor based on subjects' efficacy responses during the trial.), Cohort C (histologically or cytologically confirmed gastric cancer (including gastroesophageal junction adenocarcinoma), failed or intolerant to standard treatment, c-MET positive. Investigators may adjust enrollment criteria after communicating with the sponsor based on subjects' efficacy responses during the trial.), Cohort D (histologically or cytologically confirmed liver cancer and cholangiocarcinoma, failed or intolerant to standard treatment, c-MET positive. Investigators may adjust enrollment criteria after communicating with the sponsor based on subjects' efficacy responses during the trial.), Cohort E(histologically or cytologically confirmed pancreatic cancer, failed or intolerant to standard treatment, c-MET positive.Investigators may adjust enrollment criteria after communicating with the sponsor based on subjects' efficacy responses during the trial.), Cohort F(histologically or cytologically confirmed renal cancer, failed or intolerant to standard treatment, c-MET positive. Investigators may adjust enrollment criteria after communicating with the sponsor based on subjects' efficacy responses during the trial.) or other sensitive tumor types identified in phase Ia trial.
   * Each cohort of participants had at least one measurable lesion that met the criteria of RECIST v1.1.
6. Recovered from toxic effects of previous last treatment before the first dose (CTCAE ≤ Grade 1, except for special cases such as alopecia and hyperpigmentation); in addition, investigators judge that the corresponding AE has no safety risks.
7. Systolic blood pressure ≤ 160 mmHg, diastolic blood pressure ≤ 100 mmHg, and no changes in antihypertensive drugs and dosages within 7 days before the first dose.
8. Organ and bone marrow function must meet the following requirements:

   * Bone marrow: Absolute neutrophil count (ANC) ≥ 1.5×10⁹/L, platelet count ≥ 75×10⁹/L, hemoglobin ≥ 90 g/L; no blood transfusion or biologic response modifier (e.g., granulocyte colony-stimulating factor, erythropoietin, interleukin-11, etc.) treatment within 14 days before the first dose.
   * Liver function: No history of cirrhosis (i.e., no decompensated cirrhosis Child-Pugh Class B or C). For subjects without liver metastasis: serum total bilirubin (TBIL) ≤ 1.5×upper limit of normal (ULN) (≤ 2.0×ULN for Gilbert syndrome), alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 2.5×ULN. For subjects with liver metastasis or liver cancer: TBIL ≤ 2.5×ULN, ALT and AST ≤ 5×ULN.
   * Renal function: Creatinine clearance rate ≥ 50 mL/min (Cockcroft-Gault formula) or serum creatinine < 1.5×ULN; urine protein qualitative ≤ 1+. If urine protein qualitative ≥ 2+, 24-hour urine protein quantitative test is required; investigators make enrollment judgment based on test results.
   * Coagulation function: Prothrombin time (PT) ≤ 1.5×ULN; international normalized ratio (INR) ≤ 1.5×ULN, and activated partial thromboplastin time (APTT) ≤ 1.5×ULN. (INR < 2.5×ULN for subjects receiving anticoagulant therapy)
9. Female subjects of childbearing age must undergo serum pregnancy test within 7 days before the start of study drug administration, with negative results; and agree to use a medically approved highly effective contraceptive method (e.g., intrauterine device, contraceptive pills, or condoms) during the study and within 3 months after the last dose of study drug. Male subjects whose partners are of childbearing age must agree to use effective contraception during the study and within 3 months after the last dose of study drug. Lactating females must agree to discontinue breastfeeding during the study and within 3 months after the last dose of study drug.
10. Phase Ib trial: Meet any of the following conditions:

    * Previously confirmed c-MET positive; lung cancer cohort requires EGFR wild-type.
    * After collecting subjects' tumor tissue samples, confirmed c-MET positive by central laboratory testing. Requirements for subjects to provide tumor samples: paraffin blocks within 2 years; paraffin-embedded sections within 6 months (at least 5 slices), or fresh tissue, etc.; tumor cell proportion in samples ≥ 20%. (If tumor samples exceed the above time requirements, communication with the sponsor is allowed to determine acceptability)
    * Definition of c-MET positive: IHC ≥ 2+; or FISH amplification (GCN ≥ 5).

Exclusion Criteria:

1. Previous or current history of other types of malignant tumors, except for the following situations:

   * Curatively treated basal cell carcinoma of the skin, superficial bladder cancer, squamous cell carcinoma of the skin, carcinoma in situ of the cervix, or carcinoma in situ of the breast.
   * Second primary cancer that has been cured with no recurrence within 5 years.
2. Subjects allergic to any component of the study drug or with a history of severe allergies.
3. Received any of the following treatments or drugs before the first study treatment:

   * Major surgery or severe trauma within 4 weeks before the first study drug administration (major surgery is defined as any invasive surgery involving extensive resection or opening of mesothelial barriers such as pleural cavity, peritoneal cavity, or meninges; however, tissue biopsy for diagnostic purposes is allowed. Severe trauma refers to unhealed wounds, ulcers, or fractures).
   * Traditional Chinese medicine (including proprietary Chinese medicine) with antitumor indications within 2 weeks before the first study drug administration.
   * Antitumor treatment (including chemotherapy, radiotherapy, immunotherapy, targeted therapy, biotherapy, or tumor embolization) within 2 weeks before the first dose or within 2 half-lives of the therapeutic drug (whichever is shorter).
   * Strong CYP3A4 inducers or inhibitors within 2 weeks before the first dose and for less than 5 half-lives.
   * Drugs known to significantly prolong the QT interval (e.g., Class Ia and III antiarrhythmic drugs) within 1 week before the first dose.
4. Subjects with meningeal metastasis.
5. Subjects with a history of other central nervous system (CNS) metastases or spinal cord compression; enrollment is allowed if the following conditions are met:

   * Clearly received treatment and clinically stable after discontinuing anticonvulsants and steroids for 4 weeks before the first study drug administration (clinical stability is defined as no clinical accompanying symptoms such as increased intracranial pressure or neurological symptoms within 4 weeks and imaging suggesting stable lesions within 4 weeks before the first dose).
   * For subjects with brain metastasis: Interval from whole-brain radiotherapy (WBRT) to the first study treatment administration ≥ 21 days; interval from stereotactic radiosurgery (SRS) to the first study treatment administration ≥ 7 days; or interval from surgical resection to the first study treatment administration ≥ 28 days.
6. Advanced subjects with symptomatic visceral dissemination at risk of life-threatening complications in the short term; subjects who underwent at least two puncture drainages within 4 weeks before the first dose; or subjects who underwent one puncture drainage but with unstable pleural effusion, peritoneal effusion, or pericardial effusion.
7. Cardiovascular diseases meeting any of the following within 6 months before screening:

   * Congestive heart failure with New York Heart Association (NYHA) Class ≥ III.
   * Left ventricular ejection fraction (LVEF) < 50%.
   * Severe arrhythmia requiring drug treatment.
   * QTcF (Fridericia formula) > 450 milliseconds, or risk factors for torsades de pointes (TdP), such as clinically significant hypokalemia (e.g., CTCAE severity ≥ Grade 3 or requiring intravenous treatment) judged by investigators, family history of long QT syndrome, or family history of arrhythmia (e.g., Wolff-Parkinson-White syndrome)
   * Myocardial infarction, severe/unstable angina pectoris within 6 months before administration.
   * History of Grade ≥ 3 thromboembolic events within the past 2 years, or receiving thrombolysis due to high thrombosis risk.
8. Presence of other serious diseases, including liver disease, kidney disease, neuropsychiatric disease, endocrine disease, hematological disease, and immune system disease, which investigators judge will affect participation in the study.
9. Enlargement of the thyroid or parathyroid gland.
10. Current acute lung disease, interstitial lung disease or pneumonia, pulmonary fibrosis, acute pulmonary disease, etc., excluding local interstitial pneumonia induced by radiotherapy.
11. Subjects with clear gastrointestinal bleeding tendency, including the following situations: History of melena or hematemesis within 2 months; investigators judge that massive gastrointestinal bleeding may occur.
12. Previous or current history of Grade ≥ 3 gastrointestinal perforation or visceral fistula.
13. Adverse events from previous treatment failed to recover to ≤ Grade 1, except for alopecia, clinically insignificant abnormal laboratory findings related to the disease, hypothyroidism stabilized by hormone replacement therapy, and other toxicities with no safety risks judged by investigators.
14. Evidence of active infection:

    * Hepatitis B (simultaneous positivity for HBsAg and HBV-DNA ≥ 2000 IU/ml).
    * Hepatitis C (simultaneous positivity for HCV antibody (HCV-Ab) and HCV-RNA above the lower limit of detection of the analytical method).
    * Systemic anti-infective treatment for ≥ 7 days within 4 weeks before the first dose, or unexplained fever > 38.5℃ during screening/before the first dose (fever caused by tumors is allowed as judged by investigators).
    * Active pulmonary tuberculosis infection detected by medical history or CT examination, or history of active pulmonary tuberculosis infection within 1 year before enrollment, or history of active pulmonary tuberculosis infection more than 1 year ago without regular treatment.
15. Positive for human immunodeficiency virus (HIV RNA) or Treponema pallidum antibody.
16. Previous clear history of neurological or psychiatric disorders, including epilepsy or dementia.
17. Received any investigational drug within 4 weeks before the first dose, or concurrently participating in another clinical study (exceptions: subjects participating in observational, non-interventional clinical studies, or in the follow-up period of interventional clinical studies; or the last study drug administration was more than 5 half-lives ago).
18. Subjects judged by investigators as unsuitable for inclusion in the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2028-03-01 (Estimated); Study Completion 2029-03-01 (Estimated)

PRIMARY OUTCOMES:
Phase Ia: Dose-Limiting Toxicity (DLT) | From enrollment to the end of cycle 1,cycle 1 has 28 days.
  Continuously monitor safety; record toxic events meeting predefined criteria (NCI-CTCAE V5.0 Grade 3/4 non-hematological toxicity, Grade 4 hematological toxicity >7 days, etc.). Include subjects with ≥75% planned dose or withdrawal due to DLT; causality confirmed by investigators.
Phase Ia: Maximum Tolerated Dose (MTD) | Through the completion of cycle 1 for all phase Ia subjects,an average of 1 year.
  Adopt accelerated titration + "3+3" design; calculate DLT incidence per dose group. MTD is the maximum dose with ≤1/6 DLT cases, requiring at least 6 evaluable subjects.
Phase Ia: Assessment of safety and toxicity profile | From enrollment until the 28 days after the last study dose.
  Number of participants who experienced AEs, SAEs, and changes in physical examination, vital signs, ECOG score,imaging examination, laboratory tests, and 12-lead electrocardiogram, etc.
Phase Ib: Objective Response Rate (ORR) | From enrollment to the date of first documented progression or death due to any cause, whichever came first (up to approximately 2 years).
  Evaluate by contrast-enhanced CT/MRI (RECIST v1.1; mRECIST for hepatocellular carcinoma). ORR = proportion of subjects with CR+PR (first response confirmed after 4 weeks).

SECONDARY OUTCOMES:
Phase Ia: Objective Response Rate (ORR) | From enrollment to the date of first documented progression or death due to any cause, whichever came first (up to approximately 2 years).
  Assessed in subjects with measurable lesions at baseline per Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1. Proportion of subjects achieving CR or PR after treatment.
Phase Ia and Phase Ib: Disease Control Rate (DCR) | From enrollment to the date of first documented progression or death due to any cause, whichever came first (up to approximately 2 years).
  Assessed per RECIST v1.1. Proportion of subjects achieving CR, PR, or Stable Disease (SD) after treatment.
Phase Ia and Phase Ib: Duration of Response (DOR) | From enrollment to the date of first documented progression or death due to any cause, whichever came first (up to approximately 2 years).
  Time from the first documentation of objective response (CR/PR) to the first occurrence of disease progression or death from any cause.
Phase Ia and Phase Ib: Progression-Free Survival (PFS) | From enrollment to the date of first documented progression or death due to any cause, whichever came first (up to approximately 2 years).
  Time from the start of treatment to the first occurrence of disease progression or death from any cause.
Phase Ia and Phase Ib: Overall Survival (OS) | From enrollment to the date of death due to any cause (up to approximately 2 years).
  Time from the start of treatment to death from any cause.
Phase Ia and Phase Ib: Terminal Phase Half-life (t1/2 ) | From enrollment to the end of cycle 1,cycle 1 has 28 days.
  Evaluate drug concentration-time data by individual subject for single or repeated dosing of TPD3310.
Phase Ia and Phase Ib: Maximum plasma concentration (Cmax) | From enrollment to the end of cycle 1,cycle 1 has 28 days.
  Evaluate drug concentration-time data by individual subject for single or repeated dosing of TPD3310.
Phase Ia and Phase Ib: Time to reach Cmax (tmax) | From enrollment to the end of cycle 1,cycle 1 has 28 days.
  Evaluate drug concentration-time data by individual subject for single or repeated dosing of TPD3310.
Phase Ia and Phase Ib: Area Under the Curve (AUC) | From enrollment to the end of cycle 1,cycle 1 has 28 days.
  Evaluate drug concentration-time data by individual subject for single or repeated dosing of TPD3310.
Phase Ia and Phase Ib: Apparent Volume of Distribution (Vz/F) | From enrollment to the end of cycle 1,cycle 1 has 28 days.
  Evaluate drug concentration-time data by individual subject for single or repeated dosing of TPD3310.
Phase Ia and Phase Ib: Apparent Clearance Rate (CL/F) | From enrollment to the end of cycle 1,cycle 1 has 28 days.
  Evaluate drug concentration-time data by individual subject for single or repeated dosing of TPD3310.
Phase Ib: Assessment of safety and toxicity profile | From enrollment until the 28 days after the last study dose.
  Number of participants who experienced AEs, SAEs, and changes in physical examination, vital signs, ECOG score,imaging examination, laboratory tests, and 12-lead electrocardiogram, etc.

CONTACTS AND LOCATIONS:
Locations (1):
- Cancer Hospital Chinese Academy of Medical Sciences, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No